CLINICAL TRIAL: NCT03165123
Title: Effect of Adding Azithromycin to Dexamethasone in Preventing Post-operative Nausea and Vomiting in Caesarean Section Under Spinal Anesthesia With Spinal Opiate.
Brief Title: Effect of Using Azithromycin Versus Placebo With Dexamethasone in Prevention of Post-spinal Nausea and Vomiting.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, KAGergis, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABCD
Record Dates: First submitted 2017-05-15; First posted 2017-05-24 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Post-operative Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): The patients will receive oral placebo tablet, one hour before induction of anesthesia and 5 mg Intra-venous dexamethasone within 1-2 minutes after the umbilical cord is clamped.
  Interventions: Drug: Intravenous dexamethasone
- Azithromycin group (Active Comparator): The patients will receive 250 mg oral Azithromycin tablet, one hour before induction of anesthesia and 5 mg Intra-venous dexamethasone within 1-2 minutes after the umbilical cord is clamped.
  Interventions: Drug: Oral Azithromycin tablet; Drug: Intravenous dexamethasone

INTERVENTIONS:
Drug: Oral Azithromycin tablet — Oral azithromycin tablet will be given one hour before induction of anaesthesia.
  Arms: Azithromycin group
Drug: Intravenous dexamethasone — 5 mg of intravenous dexamethasone is given within one to two minutes after the umbilical cord is clamped.

SUMMARY:
Postoperative nausea and vomiting is defined as any nausea, retching, or vomiting occurring during the first 24-48 h after surgery in inpatients. Postoperative nausea and vomiting is one of the most common causes of patient dissatisfaction after anesthesia, with reported incidences of 30% in all post-surgical patients and up to 80% in high-risk patients. In addition, postoperative nausea and vomiting is regularly rated in preoperative surveys, as the anesthesia outcome the patient would most like to avoid. While suture dehiscence, aspiration of gastric contents, esophageal rupture, and other serious complications associated with postoperative nausea and vomiting are rare, nausea and vomiting is still an unpleasant and all-too-common postoperative morbidity that can delay patient discharge from the post-anesthesia care unit and increase unanticipated hospital admissions in outpatients.

DETAILED DESCRIPTION:
There are many well-established risk factors for Postoperative nausea and vomiting which are classified in two classes:

A) Patient related risk factors:

1. Female gender is consistently the strongest risk factor for postoperative nausea and vomiting, female patient are three times more likely than men to suffer from postoperative nausea and vomiting.
2. For adult patient, age is a statistically, though not clinically, relevant risk factor, with the incidence of postoperative nausea and vomiting decreasing as patients age. For pediatric patients, however, age increases the risk of post-operative vomiting , such that children older than 3 years have been shown to have an increased risk of post-operative vomiting compared with children younger than 3 years.
3. Obesity is a strong risk factor for postoperative nausea and vomiting : patients with body mass index more than 30 have the double risk of postoperative nausea and vomiting.
4. Non-smoking status roughly doubles the patient's risk of postoperative nausea and vomiting. The specific mechanism underlying smoking's protective effect is unknown, but one of the most commonly believed theories is that polycyclic aromatic hydrocarbons in cigarette smoke induce cytochrome P450 enzyme which increase the metabolism of emetogenic volatile anesthetics.
5. History of gastrointestinal disease as gastritis, gastric ulcer or duodenal ulcer increases the risk for postoperative nausea and vomiting.
6. History of motion sickness, Meniere's disease or previous postoperative nausea and vomiting indicates a general susceptibility to postoperative nausea and vomiting.

B) Anesthesia related risk factors:

1. The use of volatile anesthetics is associated with a two-fold increase in the risk of postoperative nausea and vomiting , with risk increasing in a dose dependent manner.
2. Intraoperative and postoperative opioid use increases the risk of postoperative nausea and vomiting in a dose dependent manner by the mechanism of reducing muscle tone and peristaltic activity, thereby delaying gastric emptying, inducing distention, and triggering the vomiting reflex.
3. The duration of anesthesia can help predict the patient's risk of postoperative nausea and vomiting, since the duration of anesthesia describes the patient's exposure to emetogenic stimuli like volatile anesthetics and intraoperative opioids.

There are two lines of anti-emetic drugs used to treat postoperative nausea and vomiting :

The first line is classified into three classes: serotonin antagonists (e.g. ondansetron), corticosteroids (e.g. dexamethasone), and dopamine antagonists (e.g. droperidol) have similar efficacy against postoperative nausea and vomiting , with a relative risk reduction of ~25%. Moreover, they act independently and when used in combination, have additive effects.

Dexamethasone can be effective in preventing postoperative nausea and vomiting in adults and children. Compared with other operative medications, dexamethasone has equal or even better efficacy in reducing the incidence of Postoperative nausea and vomiting and has the advantages of low cost and longer effectiveness as well. The mechanism of the antiemetic action of dexamethasone is still not clearly known. Glucocorticoids receptors are found in nucleus of the solitary tract, the raphe nucleus and the area postrema and all are associated with regulating nausea and vomiting. Dexamethasone may affect postoperative nausea and vomiting by modulating neurotransmission or receptor density in these nuclei. Clinically, dexamethasone as a preventive drug against postoperative nausea and vomiting has not caused fatal outcome; therefore, it is generally considered to be an effective and safe anti-emetic. Nevertheless, its use in this regard may lead to adverse effects, principally postoperative hyperglycemia and infection.

The second line is characterized by less favorable side effect profiles or limited evidence of efficacy: Metoclopramide is a widely used D2 antagonist. Contrary to popular belief, the 10 mg dose has no effect on post-operative nausea and vomiting, but 25-50 mg has similar efficacy compared with other anti-emetics. Metoclopramide use has been associated with extrapyramidal and sedative side-effects. Dimenhydrinate is an antihistamine like promethazine and cyclizine. There are few randomized controlled trials investigating its use for postoperative nausea and vomiting , and the drug is associated with a significant rate of side-effects like sedation, dry mouth, visual disturbance, and urinary retention.

Azithromycin , one of macrolides, was introduced in the 1950s and after years of clinical experience it still remains a commonly relied upon antibiotic but the function of erythromycin as a prokinetic agent has also been investigated recently for a range of gastrointestinal motility disorders and more recently within the context of critically ill patients. Azithromycin has a gastrointestinal motility stimulating effect; it has been known for over 20 years that they act as a motilin receptor agonist in the gut and gallbladder stimulating enteric nerves and smooth muscle and triggering a phase of the migrating myoelectric complex. The antral motor effects of erythromycin A in humans are mediated via different pathways. The induction of a premature activity is mediated through activation of an intrinsic cholinergic pathway, while the induction of enhanced antral contractile activity may be mediated via a pathway potentially involving activation of non muscular receptor. Different doses of azithromycin may have different effects - as suggested in studies in patients with diabetic gastro-paresis.

Forty mg azithromycin elicited a premature phase 3 complex that started in the stomach and migrated to the small intestine, while doses of 200 and 350 mg erythromycin A elicited a burst of antral phase-3-like contractions that did not migrate to the small intestine, but were followed by a prolonged period of antral contractile activity.

ELIGIBILITY:
Inclusion Criteria: 1- women classified according to American Society of anaesthesiologists grade I between the ages 18 to 38 years scheduled for elective Caesarean Section under spinal anesthesia who are normal healthy women, non smokers, no or minimal alcohol use.

2- women classified as American Society of Anaesthesiologists grade Il between the ages 18 to 38 years scheduled for elective Caesarean Section under spinal anesthesia who are women with mild systemic disease without functional limitations as current smokers, social alcohol drinker, pregnant, women with body mass index between 30 and 40, women with well-controlled diabetas, hypertension or mild lung diseases.

Exclusion Criteria:

1. Women who has obstetric complications.
2. Women with evidence of foetal compromise.
3. Patients who have gastro-intestinal diseases.
4. Patients who administrated anti-emetic medication in the previous 24 hours before operation.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Direct questionnaire of the patients about their nausea and/or vomiting | The first 24 hours after surgery
  1. Did you experience nausea during the first 24 hours after your surgery?
     1. yes
     2. no [if no, please skip to question 5]
  2. How long did the nausea last? ....... hours.
  3. How would you describe the nausea at its worst?
     1. mild
     2. moderate
     3. severe
     4. intolerable
  4. How many times you felt nauseated? ......
  5. Did you experience vomiting during the first 24 hours after your surgery?
     1. yes
     2. no [ if no, please skip the next part of the questionnaire]
  6. How would you describe the vomiting at its worst?
     1. mild
     2. moderate
     3. severe
     4. intolerable
  7. How many times you vomited during the first 24 hours after your surgery? .......
  8. Estimate the amount of the vomiting?
     1. small amount
     2. moderate amount
     3. large amount

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Aleem M, Osman A, Morsy K. Effect of coadministration of dexamethasone with intrathecal morphine on postoperative outcomes after cesarean delivery. Int J Gynaecol Obstet. 2012 Feb;116(2):158-61. doi: 10.1016/j.ijgo.2011.10.002. Epub 2011 Oct 26. PMID 22036059
- [Result] Rea E, Husbands E. Erythromycin: prophylaxis against recurrent small bowel obstruction. BMJ Support Palliat Care. 2017 Sep;7(3):261-263. doi: 10.1136/bmjspcare-2017-001343. Epub 2017 Mar 29. PMID 28356304
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866